CLINICAL TRIAL: NCT00368212
Title: Treating Refractory Symptoms in Primary Care (Hypochondriasis: Diagnosis, Description and Medical Care)
Brief Title: Integrated Treatment Program for Hypochondriasis in Primary Care Settings
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Arthur Joseph Barsky III,M.D., principal investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH040487 (NIH); R01MH040487 (NIH); DSIR 82-SEPC
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Hypochondriasis; Somatoform Disorders
Keywords: Somatization; Refractory Symptoms
MeSH Terms: conditions — Hypochondriasis; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive psychoeducational counseling (termed "health care counseling")
  Interventions: Behavioral: Psychoeducational counseling
- 2 (Active Comparator): Participants will receive relaxation response training
  Interventions: Behavioral: Relaxation response training

INTERVENTIONS:
Behavioral: Relaxation response training — The control treatment is relaxation training or attention control. This will be taught in three, 1-hour sessions with a trained therapist.
  Other Names: Relaxation and Stress Reduction
  Arms: 2
Behavioral: Psychoeducational counseling — Patients will receive five sessions of psychoeducational counseling from the nurse who works with the primary care physicians. Patients who are interested in continuing treatment or who have not responded to this first treatment step will then be referred for the second step, cognitive behavioral therapy (CBT), for more intensive treatment.
  Other Names: Educational Counseling
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of an integrated three-part treatment program in improving the quality of care and treatment outcomes of people with hypochondriasis in primary care settings.

DETAILED DESCRIPTION:
Hypochondriasis, which is classified as a type of somatoform disorder, is one of the most difficult psychiatric disorders to treat. It is prevalent in primary care settings, and is a major source of suffering for patients and frustration for physicians. People with hypochondriasis tend to become preoccupied with the fear of having a serious disease, despite appropriate medical evaluations and reassurance that indicate otherwise. The disorder usually occurs in episodes lasting from months to years, separated by equally long periods of quiescence. Existing strategies for treating hypochondriasis include psychotherapy, medication treatment, and alternative treatments, such as exercise and electroconvulsive therapy. An effective treatment program should target the needs of both patients and physicians, as well as the structure of the delivery system. Components of such a program have been developed, but have not yet been integrated and tested in a clinical setting. This study will evaluate the effectiveness of an integrated three-part treatment program in improving hypochondriasis treatment and quality of care outcome in primary care settings.

Participants in this 6-month, single-blind study will first undergo baseline assessments. They will then be randomly assigned to partake in either the three-part treatment program or relaxation response training, in which patients are taught to use muscle relaxation techniques to reduce stress. Over the course of the study, participants assigned to the three-part program will attend five self-scheduled, 30-minute sessions of psychoeducational counseling based on cognitive behavioral therapy principles. Sessions will focus on common hypochondriacal cognitive distortions and misunderstandings about symptoms, disease, and medical care. Additionally, the doctors and nurses at the participating hospital will undergo a training program to improve medical management of patients with hypochondriasis. The final component of the program will entail implementing an enhanced role for nurse practitioners to collaborate with primary care physicians in caring for patients with hypochondriasis. Participants assigned to relaxation response training will attend three self-scheduled, 1-hour sessions over the course of the study. They will be provided with an explanation of the physical effects of stress on the body and the purposes of progressive muscle relaxation training. They will then learn a relaxation technique through direct instruction, and will practice between sessions. Participants will also use a 20-minute audio tape to practice once a day, 5 to 7 days a week between clinic visits. All participants will attend self-scheduled follow-up visits 6 and 12 months following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has received primary medical care at Harvard Vanguard Medical Associates (HVMA) for at least 12 months prior to study entry
* Expects to continue receiving care from the current primary care physician for at least the next 12 months
* Meets requirement for average hypochondriasis screening score
* Able to speak and read English
* Falls within the top 20% of utilizers of health care services in the HVMA system over the past year
* Has attended no more than one visit to any specialist over the year prior to study entry

Exclusion Criteria:

* Psychiatric illness (e.g., psychosis, dementia, suicidal ideation)
* Somatoform pain disorder or currently receiving treatment for somatoform pain disorder (e.g., relaxation training)
* History of alcohol or substance abuse or dependence within the 12 months prior to study entry
* Terminal medical illness or major medical illness expected to worsen significantly over the next year
* Ongoing symptom-contingent litigation against HVMA
* Monetary compensation for medical disability

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2005-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Whitely Index | Measured immediately post-treatment and at Months 6 and 12 post-treatment

SECONDARY OUTCOMES:
Health Anxiety Inventory | Measured immediately post-treatment and at Months 6 and 12 post-treatment
Modified Cognitions Questionnaire | Measured immediately post-treatment and at Months 6 and 12 post-treatment
Somatic Symptom Inventory | Measured immediately post-treatment and at Months 6 and 12 post-treatment
Functional Status Questionnaire | Measured immediately post-treatment and at Months 6 and 12 post-treatment
Client Satisfaction Index | Measured immediately post-treatment and at Months 6 and 12 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arthrur J. Barsky, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Harvard Vanguard Medical Associates, Cambridge, Massachusetts

REFERENCES:
- [Derived] Barsky AJ, Ahern DK, Bauer MR, Nolido N, Orav EJ. A randomized trial of treatments for high-utilizing somatizing patients. J Gen Intern Med. 2013 Nov;28(11):1396-404. doi: 10.1007/s11606-013-2392-6. Epub 2013 Mar 14. PMID 23494213